CLINICAL TRIAL: NCT03502343
Title: Efficacy and Safety of Modified Nab-Paclitaxel Plus Gemcitabine Chemotherapy for Metastatic Pancreatic Cancer: A Single-arm Phase II Clinical Trial
Brief Title: Efficacy and Safety of Modified Nab-Paclitaxel Plus Gemcitabine Chemotherapy for Metastatic Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0840
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic cancer; Metastatic; Modified; Gemcitabine; nab-Paclitaxel
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Modified Gemcitabine plus nab-Paclitaxel (Experimental): The intervention group
  Interventions: Drug: Modified Gemcitabine plus nab-Paclitaxel Combination Chemotherapy

INTERVENTIONS:
Drug: Modified Gemcitabine plus nab-Paclitaxel Combination Chemotherapy — All patients will receive slow (over 30-40 minutes) intravenous administration of nab-paclitaxel (125 mg/m2) on days 1 and 15, and gemcitabine (1000 mg/m2) on days 1, 8, and 15 of a 28- day cycle (every 4 weeks). Treatment will discontinue if disease progression or intolerable toxicity is observed, if the patient withdraws from the study, or at the physician's discretion.
  Dose reduction of the chemotherapeutic agent and/or delay of administration is allowed if serious treatment-related AEs occur, according to specified guideline in study protocol (Level 1: 100% -> 80%; Level 2: 80% -> 60%). If dose reduction is needed more than Level 2, the patient will be dropped from the trial.

SUMMARY:
Recently, a retrospective study reported the efficacy and safety of modified gemcitabine plus nab-paclitaxel (GnP), which were administered biweekly (on days 1 and 15). With 79 patients of metastatic pancreatic cancer, this study reported similar efficacy and improved toxicity profile compared with standard dose GnP (OS 10 months, PFS 5.4 months, Grade ≥3 Neutropenia 19%, Grade ≥3 sensory neuropathy 1.6%). Also, several studies reported that dose reduction of nab-paclitaxel in breast or pancreatic cancer treatment was not related of decreased survival, or related with prolonged survival and increased treatment exposure. However, this finding need to be evaluated in prospective clinical trial.

This phase II trial will evaluate the efficacy and safety of modified GnP, which omit the day 8 administration of nab-paclitaxel, in metastatic pancreatic cancer.

DETAILED DESCRIPTION:
Gemcitabine-based combination therapy have been used to prolong survival for patient with pancreatic cancer. In early 2010s, gemcitabine plus nab-paclitaxel (GnP) combination regimen have been introduced based on the results of randomized phase III clinical trial that showed survival benefit than gemcitabine monotherapy. Nab-paclitaxel is a nanoparticle albumin-bound paclitaxel that showed anti-tumor activity as well as synergistic effect in combination with gemcitabine.

In the Metastatic Pancreatic Adenocarcinoma Clinical Trial (MPACT), the maximal tolerated nab-paclitaxel dose (125 mg/m2) was administrated with 1000 mg/m2 of gemcitabine, on days 1, 8 and 15 for 4 weeks cycle. This combination therapy showed favorable treatment response, but notable severe adverse events were also reported. Grade 3 or higher neuropathy and neutropenia occurred in 17% and 38% of patients, respectively. Also, dose reduction was required in approximately half of the patients.

Recently, a retrospective study reported the efficacy and safety of modified GnP, which were administered biweekly (on days 1 and 15). With 79 patients of metastatic pancreatic cancer, this study reported similar efficacy and improved toxicity profile compared with standard dose GnP (OS 10 months, PFS 5.4 months, Grade ≥3 Neutropenia 19%, Grade ≥3 sensory neuropathy 1.6%). Also, several studies reported that dose reduction of nab-paclitaxel in breast or pancreatic cancer treatment was not related of decreased survival, or related with prolonged survival and increased treatment exposure. However, this finding need to be evaluated in prospective clinical trial.

This phase II trial will evaluate the efficacy and safety of modified GnP, which omit the day 8 administration of nab-paclitaxel, in metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically confirmed pancreatic adenocarcinoma
* Coexisting extrapancreatic distant metastasis
* Older than 19 years old
* Measurable primary tumor in pancreas on imaging study at the time of diagnosis, according to the RECIST criteria

Exclusion Criteria:

* Previous history of palliative systemic chemotherapy due to pancreatic cancer
* Existence of active malignancy of other organ which diagnosed in last five years (except the squamous cell carcinoma or basal cell tumor of skin)
* Existence of life-threatening co-morbidity
* Poor performance state (ECOG ≥2)
* Suspected severe bone marrow suppression (Neutrophil count< 1,500/mm3, Hemoglobin< 9 g/dL, Platelet count< 75,000/mm3)
* Suspected severe liver dysfunction (Total bilirubin or Prothrombin Time > 1.5 times of upper normal range) or renal dysfunction (estimated GFR < 50/ml/min/1.73 m²)
* Pre-existence of ≥grade 2 peripheral sensory neuropathy
* Existence of brain metastasis or meningeal carcinomatosis
* Patient with pregnancy or ongoing breast feeding
* Do not agree with the informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Every 8 weeks until dropout up to 104 weeks
  To evaluate treatment efficacy, computed tomography scan, magnetic resonance imaging, or 18F-fluorodeoxyglucose-positron emission tomography (18F-FDGPET) scan will be performed every 8 weeks. Treatment responses according to the RECIST criteria will be reported by designated radiologists and final disease assessment will be independently made by the attending physician. The proportion of patients with the best response of complete response (CR), partial response (PR) is defined as objective response rate.
Disease control rate | Every 8 weeks until dropout up to 104 weeks
  To evaluate treatment efficacy, computed tomography scan, magnetic resonance imaging, or 18F-fluorodeoxyglucose-positron emission tomography (18F-FDGPET) scan will be performed every 8 weeks. Disease control rate is defined as the proportion of patients with the best response of CR, PR and stable disease.

SECONDARY OUTCOMES:
Overall survival | Every 8 weeks from date of drug administration until the date of patient's death, loss of follow-up, or end of the trial up to 104 weeks
  The overall survival is defined as from the date of enrollment to the date of the last follow-up or death of all causes. In case of loss of follow-up, the censoring date will be the day on which the survival is confirmed before follow-up loss.
Progression-free survival | Every 8 weeks from date of drug administration until the date of patient's death, loss of follow-up, or end of the trial up to 104 weeks
  The progression free survival is defined as from the date of treatment initiation to the date of the event. The event is defined as the date of disease progression or patient's death, which occured first.
  In case of loss of follow-up, the censoring date will be the day on which the survival is confirmed before follow-up loss.
Adverse event | Until dropout from the trial up to 104 weeks
  Adverse events will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.03) before each cycle until study dropout.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Von Hoff DD, Ervin T, Arena FP, Chiorean EG, Infante J, Moore M, Seay T, Tjulandin SA, Ma WW, Saleh MN, Harris M, Reni M, Dowden S, Laheru D, Bahary N, Ramanathan RK, Tabernero J, Hidalgo M, Goldstein D, Van Cutsem E, Wei X, Iglesias J, Renschler MF. Increased survival in pancreatic cancer with nab-paclitaxel plus gemcitabine. N Engl J Med. 2013 Oct 31;369(18):1691-703. doi: 10.1056/NEJMoa1304369. Epub 2013 Oct 16. PMID 24131140
- [Background] Ahn DH, Krishna K, Blazer M, Reardon J, Wei L, Wu C, Ciombor KK, Noonan AM, Mikhail S, Bekaii-Saab T. A modified regimen of biweekly gemcitabine and nab-paclitaxel in patients with metastatic pancreatic cancer is both tolerable and effective: a retrospective analysis. Ther Adv Med Oncol. 2017 Feb;9(2):75-82. doi: 10.1177/1758834016676011. Epub 2016 Nov 2. PMID 28203300
- [Background] Gradishar WJ, Krasnojon D, Cheporov S, Makhson AN, Manikhas GM, Clawson A, Bhar P, McGuire JR, Iglesias J. Phase II trial of nab-paclitaxel compared with docetaxel as first-line chemotherapy in patients with metastatic breast cancer: final analysis of overall survival. Clin Breast Cancer. 2012 Oct;12(5):313-21. doi: 10.1016/j.clbc.2012.05.001. Epub 2012 Jun 23. PMID 22728026
- [Background] Scheithauer W, Ramanathan RK, Moore M, Macarulla T, Goldstein D, Hammel P, Kunzmann V, Liu H, McGovern D, Romano A, Von Hoff DD. Dose modification and efficacy of nab-paclitaxel plus gemcitabine vs. gemcitabine for patients with metastatic pancreatic cancer: phase III MPACT trial. J Gastrointest Oncol. 2016 Jun;7(3):469-78. doi: 10.21037/jgo.2016.01.03. PMID 27284481